CLINICAL TRIAL: NCT07221773
Title: Pilot Study to Evaluate the Efficacy and Safety of Xvie (Human Amniotic Fluid Derived Nanoparticle Solution) Delivered Into the Scalp by Microneedling in Women With Self-perceived Thinning Hair
Brief Title: Pilot Study to Evaluate the Efficacy and Safety of Xvie Delivered Into the Scalp by Microneedling in Women With Self-perceived Thinning Hair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Restore Biologics Holdings, Inc. dba Xtressé (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XVIEP-2025-001
Record Dates: First submitted 2025-10-23; First posted 2025-10-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hair Thinning
Keywords: hair loss; hair thinning; Alopecia; thin hair; thinning hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Open label study evaluating safety and efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XVIE microneedling process applied to the scalp twice over a 4 month period. (Experimental): XVIE is proprietary, additive-free human amniotic fluid derived product that contains an diverse array of bioreactive molecules including growth factors, cytokines, ECM proteins, exosomes, and hyaluronic acid.
  Interventions: Other: XVIE

INTERVENTIONS:
Other: XVIE — Acellular Allogenic Human Amniotic Fluid (hAF)

SUMMARY:
The goal of this study is to determine how safe and effective it is to improve hair growth using XVIE solution applied on the scalp of women with self-perceived thinning hair.

The main aims of this trial are:

1. To confirm using photographic analysis, changes in the quality, volume, and thickness of hair.
2. To gauge patient satisfaction with hair changes and application process.

Participants who qualify will complete 5 to 6 visits after voluntary consent has been given. Participant's scalp will be numbed and the XVIE solution will be applied by microneedling. Photographs will be taken at each visit to measure changes in hair volume, thickness, and growth. Every participant will receive active treatment twice over the 4 month period.

DETAILED DESCRIPTION:
XVIE is a proprietary, additive-free Human amniotic fluid (hAF) based therapy, containing a diverse array of bioactive molecules including growth factors, cytokines, hyaluronic acid, extracellular matrix proteins, and extracellular vesicles including exosomes. Extensive research have shown the ability of Xvie components to support cellular proliferation, angiogenesis, immune regulation, and matrix remodeling which has the potential to reverse underlying cause of hair loss.

In the study, participants will be asked to complete the following:

* Provide basic personal Information
* Provide a Medical & Surgical History
* Follow study requirements to avoid certain medication and treatments
* Complete all study visits and follow-up calls
* Complete self-assessments and treatment use logs
* Allow clinical assessment and photographic documentation of treatment.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 28-65 years with self-perceived thinning hair (confirmed by an investigator).
* Ludwig Scale 1 to 2
* Fitzpatrick skin types I to VI.
* Ability and willingness to comply with the study protocol.
* Commitment to using effective contraception throughout the study if of childbearing potential.

Exclusion Criteria:

* Pregnancy, nursing, or recent initiation of hormone therapy.
* Change in other hair treatments within 3 months prior to the study.
* Known uncontrolled health conditions (e.g., poorly controlled diabetes, hypertension).
* History of hair or scalp disorders that could interfere with study results.
* History of keloid formation or poor wound healing
* History of bleeding and/or clotting disorders

Ages: 28 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex at birth
Enrollment: 15 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Within-subject increase in hair quality, volume, and thickness, assessed via Canfield HairMetrix® Phototrichogram Analysis | From enrollment to the end of treatment at 4 months
  Quantitative hair measurements calculated by analyzing the participants digital images from baseline to 4 months after multiple treatments with XVIE
Incidence of Adverse Events associated with Treatment | From first treatment until the end of treatment at 4 months.
  Collect and quantify the incidence of treatment-related adverse events and treatment-related serious adverse events that occur during the trial within 30 days of microneedling treatment.

SECONDARY OUTCOMES:
Hair Density Changes measured by SOCAi | From enrollment to the end of the study at 4 months
  Images will be captured using the the SOCAi system at baseline and Days 30, 60, 90, and 120, to evaluate hair density changes.

OTHER OUTCOMES:
Participant self-assessment of hair improvements collected via questionnaires | From enrollment to the end of study at 4 months
  Observations and changes noted in hair loss graded on scale of 0 to 4 with 0 as no change and 4 as a very severe outcome.
  Observations and changes noted in quality of life based on hair loss, with outcomes graded between extremely effected to not at all.
  Observations are based on self-assessments completed at baseline and Day 120.
Investigator assessment of changes in hair quality | From baseline to the end of the study at 4 months
  Changes noted in hair quality graded on a scale of -3 to +3, with -3 as decreased/significantly worsened, 0 indicates no change, and +3 as increased/significantly improved

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Y Rayner, MS, Study Director — Restore Biologics Holding, Inc dba Xtressé
Locations (2):
- United States (2):
  - Advanced Dermatology & Cosmetic Surgery, Maitland, Florida
  - Kindred Hair & Skin Center, Marriottsville, Maryland

IPD SHARING:
Plan to Share IPD: No